CLINICAL TRIAL: NCT00381628
Title: Use of Nasal Epithelial Cells and Blood Lymphocytes to Identify Markers for Cystic Fibrosis and Cystic Fibrosis Pulmonary Exacerbations
Brief Title: Nasal Epithelial Cells/Blood Lymphocyte Markers for Cystic Fibrosis (CF)/CF Pulmonary Exacerbations
Status: Completed | Type: Observational
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Principal Investigator, James F. Chmiel, Associate Professor of Pediatrics, University Hospitals Cleveland Medical Center
Other Study IDs: Protocol 08-06-23
Record Dates: First submitted 2006-09-27; First posted 2006-09-28 (Estimated); Results first posted 2017-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-01

CONDITIONS: Cystic Fibrosis
Keywords: Anatomy; cells; epithelial cells; blood cells; cystic fibrosis; equipment and supplies; disposable equipment; reagent kits
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Stable subjects with CF: These subjects will undergo epithelial cells and blood lymphocyte extraction. Nasal curettage will be performed to obtain nasal epithelial cells and blood will be obtained to isolate circulating lymphocytes one time from these subjects (age 15 years and above) when they are in their usual state of well-health. These cells will be studied in vitro.
  Interventions: Procedure: epithelial cells and blood lymphocyte extraction
- Exacerbating subjects with CF: These subjects will undergo epithelial cells and blood lymphocyte extraction. Nasal curettage will be performed to obtain nasal epithelial cells and blood will be obtained to isolate circulating lymphocytes one time from these subjects (age 15 years and above) at the beginning and end of treatment for a pulmonary exacerbation. These cells will be studied in vitro.
  Interventions: Procedure: epithelial cells and blood lymphocyte extraction
- Stable subjects with asthma: These subjects will undergo epithelial cells and blood lymphocyte extraction. Nasal curettage will be performed to obtain nasal epithelial cells and blood will be obtained to isolate circulating lymphocytes one time from these subjects (age 15 years and above) when they are in their usual state of well-health. These cells will be studied in vitro. This is the disease control group.
  Interventions: Procedure: epithelial cells and blood lymphocyte extraction
- Healthy volunteers: These subjects will undergo epithelial cells and blood lymphocyte extraction. Nasal curettage will be performed to obtain nasal epithelial cells and blood will be obtained to isolate circulating lymphocytes one time from these subjects (age 15 years and above) when they are in their usual state of well-health. These cells will be studied in vitro. This is the control group
  Interventions: Procedure: epithelial cells and blood lymphocyte extraction

INTERVENTIONS:
Procedure: epithelial cells and blood lymphocyte extraction — Nasal curettage will be performed from each nostril to obtain nasal epithelial cells. Venipuncture will be performed and up to 60-ml of blood will be obtained from which neutrophils will be isolated.

SUMMARY:
Study Hypothesis: We hypothesize that cellular markers from nasal epithelial cells and blood lymphocytes can serve as potential biomarkers reflect the underlying inflammatory state of the lung and will be helpful in determining the presence of a CF pulmonary exacerbation and its overall severity.

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is the most common lethal genetic disease in the US afflicting approximately 30,000 people. Chronic disease of the respiratory tract, which is responsible for early death, affects both the upper and lower airways.

We propose to utilize cells (blood lymphocytes and nasal epithelial cells) that are readily accessible and are known to express the cystic fibrosis transmembrane conductance regulator (CFTR) and therefore candidates to express markers of the downstream consequences of CFTR deficiency.

A marker that indicates the inflammatory state of the lung would be useful to identify infective/inflammatory exacerbations as opposed to worsening due to pulmonary vascular disease or simply upper airway infection. This marker might help to guide therapy for intensity and duration. Evidence in mice suggest that lymphocytes may be a driving force for inflammation in the CF lung, particularly during exacerbations, and also that human CF lymphocytes have dysfunctional production of cytokines.

Specific Aims:

To identify markers in nasal epithelial cells or blood lymphocytes that distinguish CF patients from those with functional CFTR (healthy volunteers and patients with asthma). If successful this could become a marker for CFTR correction by drugs or other systemic therapies.

To identify markers in blood lymphocytes that will identify inflammatory status (ie, distinguish an active exacerbation from return to clinical stability) in CF patients. This could become a marker for infectious exacerbations of CF airway disease.

ELIGIBILITY:
Stable CF Patients:

Inclusion Criteria:

* Male or female >= 15 years of age
* Confirmed diagnosis of CF
* Clinically stable with no evidence of acute upper respiratory tract infection or current pulmonary exacerbation within the previous month
* Ability to understand and sign a written informed consent and comply with the requirements of the study

Exclusion Criteria:

* Chronic use of a medication with anti-neutrophil or anti-inflammatory effect (ibuprofen, systemic or inhaled corticosteroids, or other immunosuppressive agents, etc
* Oxygen saturation <92% on room air
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the subject or the quality of the data

CF patients with pulmonary exacerbations:

Male of female >= 15 years of age Confirmed diagnosis of CF

Patient meets a modified definition for a pulmonary exacerbation based upon Fuchs criteria which is treated with intravenous antibiotics for any 4 of the following 12 signs or symptoms:

* Increased sputum production
* New or increased coughing up of blood
* Increased cough
* Increased dyspnea with exertion
* Malaise, fatigue or lethargy
* Anorexia or weight loss
* Fever
* Sinus pain or tenderness
* Changes in sinus discharge
* New findings on chest examination
* Decline in forced expiratory volume in 1 second (FEV1) > 10% since previous visit
* Radiographic changes indicative of pulmonary infection
* Ability to understand and sign a written informed consent and comply with the requirements of the study

Exclusion criteria for CF patients with pulmonary exacerbation:

* Concurrent use a medication with anti-neutrophil or anti-inflammatory effect within the previous 4 weeks
* Presence of a condition or abnormality that in the opinion of the investigator would compromise the safety of the subject or the quality of the data.

Inclusion Criteria - Asthma patients

* Male or female >= 15 years of age
* Physician diagnosed asthma
* Clinically stable with no evidence of acute upper or lower respiratory tract infection or current pulmonary exacerbation within the previous month

Exclusion Criteria - Asthma patients

* Chronic use of a medication with anti-neutrophil or anti-inflammatory effect within the previous 4 weeks
* Treated for an asthma exacerbation with the previous 4 weeks
* Treated with oral corticosteroids within the previous 4 weeks
* Oxygen saturation <92% on room air
* Presence of a condition or abnormality that in the opinion of the investigator would compromise the safety of the subject or the quality of the data.

Inclusion Criteria for Healthy Volunteers

* Male or female >= 18 years of age
* Free of any chronic medical condition
* Clinically stable with no evidence of acute upper or lower respiratory tract infection within the previous month
* Ability to understand and sign a written informed consent and comply with the requirements of the study

Exclusion Criteria for Healthy Volunteers

* Use of a medication with anti-neutrophil or anti-inflammatory effect within the previous 4 months
* Presence of any chronic medical condition
* Oxygen saturation <92% on room air
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the subject or the quality of the data

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Nasal epithelial cells and blood will be obtained from four groups of subjects age 15 years and older: Stable subjects with CF at baseline, Subjects with CF at the beginning and end of treatment for a pulmonary exacerbation, stable subjects with asthma, and healthy voulnteers
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2006-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James F Chmiel, MD, MPH, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- Rainbow Babies and Children's Hospital, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Stable Subjects With CF | Exacerbating Subjects With CF | Stable Subjects With Asthma | Healthy Volunteers
Started | 18 | 27 | 0 | 14
Completed | 18 | 27 | 0 | 14
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stable Subjects With CF | Exacerbating Subjects With CF | Stable Subjects With Asthma | Healthy Volunteers | Total
Number analyzed (Participants) | 18 | 27 | 0 | 14 | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 2 |  | 0 | 4
  Between 18 and 65 years | 15 | 25 |  | 14 | 54
  >=65 years | 1 | 0 |  | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 10 |  | 9 | 23
  Male | 14 | 17 |  | 5 | 36
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 27 | 0 | 14 | 59

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Blood and Sputum Samples Collected
Description: Blood and sputum samples for general science research collaborators
Time Frame: Baseline
Population: These samples were to be distributed to research collaborators and were not part of a clinical trial. These samples were not analyzed for a specific outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Stable Subjects With CF | Exacerbating Subjects With CF | Stable Subjects With Asthma | Healthy Volunteers
Number analyzed (Participants) | 18 | 27 | 0 | 14
Participants | 18 | 27 | 0 | 14

ADVERSE EVENTS:
Arm/Group | Stable Subjects With CF | Exacerbating Subjects With CF | Stable Subjects With Asthma | Healthy Volunteers
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/27 | 0/0 | 0/14
Other Adverse Events (participants affected / at risk) | 1/18 | 0/27 | 0/0 | 0/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stable Subjects With CF (N=18) | Exacerbating Subjects With CF (N=27) | Stable Subjects With Asthma (N=0) | Healthy Volunteers (N=14)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No